CLINICAL TRIAL: NCT03717116
Title: Early Prediction of Hypocalcemia After Thyroidectomy Using Postoperative Second Hour Parathormone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Selen Soylu, MD, MD, Istanbul University
Other Study IDs: 83045809-604.01.02, A-01
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hypocalcemia, Postoperative Parathormone
Keywords: hypocalcemia, parathormone, bone density
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — blood samples for biochemical evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control-normocalcemia group
  Interventions: Diagnostic Test: parathormone level
- hypocalcemia group
  Interventions: Diagnostic Test: parathormone level

INTERVENTIONS:
Diagnostic Test: parathormone level — From the patients, blood will be taken preoperatively and postoperatively.
  Other Names: calcium level

SUMMARY:
Hypocalcemia is the most frequent complication in thyroid surgeries. Diagnosing this complication earlier will reduce longer hospital stay and will lead to an earlier intervention. The purpose of the study is to evaluate postoperative second hour parathyroid hormone measurement as a predictor for early stage hypocalcemia.

ELIGIBILITY:
Inclusion Criteria:

* patients with multinodular goiter, Graves, fine needle aspiartion biopsy with Bethesda 3-4 undergoing total thyroidectomy

Exclusion Criteria:

* pregnant women
* patients with thyroid cancer or previous neck dissection

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients with multinodular goiter, Graves, fine needle aspiartion biopsy with Bethesda 3-4 undergoing total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative parathormone level | postoperative 2. hour

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided